CLINICAL TRIAL: NCT02014636
Title: A Phase I/II Study to Assess the Safety and Efficacy of Pazopanib and MK 3475 in Patients With Advanced Renal Cell Carcinoma
Brief Title: Safety and Efficacy Study of Pazopanib and MK 3475 in Advanced Renal Cell Carcinoma (RCC; KEYNOTE-018)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200249; KEYNOTE-018 (Other: Merck); PZP034A2101 (Other: Novartis)
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Carcinoma, Renal Cell
Keywords: Pazopanib (GW786034); MK 3475; Renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Part 1 is a dose escalation phase in which subjects will receive pazopanib orally and the MK 3475 intravenously. Subjects will be evaluated for a minimum of 8 weeks before the next dose level cohort is enrolled.
  Interventions: Drug: Pazopanib; Drug: MK-3475
- Part 2 (Experimental): Part 2 is a randomized phase in which subjects will be enrolled in each treatment arm:
  Pazopanib monotherapy Pazopanib+MK-3475 MK-3475 monotherapy
  Interventions: Drug: Pazopanib; Drug: MK-3475

INTERVENTIONS:
Drug: Pazopanib — Pazopanib is an orally administered 200 mg tablet available in the dose range of 400 to 800 mg
Drug: MK-3475 — MK 3475 is an intravenously administered 100 mg/ 4mL solution available in the potential dose range of 1 to 10 mg/kg.

SUMMARY:
This is an open-label, 2 part study of pazopanib and/or MK 3475 in treatment naïve subjects with advanced RCC. Part 1 consists of a Phase I dose escalation of pazopanib + MK 3475 followed by an expansion cohort to determine the maximum tolerated regimen and the recommended Phase II dose. Part 2 is a randomized 3-arm Phase II study to evaluate the clinical efficacy and safety of pazopanib + MK 3475 as compared to single-agent pazopanib and single-agent MK 3475. The objectives of this Phase I/II study are to test the safety and tolerability of pazopanib in combination with MK 3475, and study the clinical efficacy of pazopanib in combination with MK 3475 in subjects with advanced RCC as compared with single-agent pazopanib and single-agent MK 3475.

Following the Urgent Safety Measure (USM) released on February 09, 2017, the phase II (Part 2) portion of this study will not commence.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up
* Diagnosis of locally advanced or metastatic RCC that is predominantly clear cell histology
* Must have measurable disease
* Subject has received no prior systemic therapy
* A woman is eligible to participate in the study if she is of Non-childbearing potential, has a negative serum pregnancy test within 7 days of the first dose of study treatment, not lactating, and agrees to use adequate contraception during the study until at least 120 days after the last dose of investigational product
* Eastern Cooperative Oncology Group performance status 0 or 1
* Adequate organ function as defined in the protocol
* Left ventricular ejection fraction >= lower limit of normal as assessed by echocardiogram or multigated acquisition scan
* In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Subject has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents
* Subject is currently participating or has participated in a study of an investigational agent or using an investigational device within 30 days of the first dose of study treatment
* Subject is expected to require any other form of systemic or localized antineoplastic therapy while on study
* Subject is on any systemic steroid therapy, within one week before the planned date for first dose of study treatment. Subject is on any other form of immunosuppressive medication
* Subject has a history of a malignancy (other than the disease under treatment in the study) within 5 years before first study treatment administration
* Central nervous system metastasis
* Unable to swallow and retain orally administered medication
* Subject has interstitial lung disease or a history of pneumonitis
* Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other Gastrointestinal conditions with increased risk of perforation; history of abdominal fistula, GI perforation, or intra-abdominal abscess within 4 weeks before beginning study treatment
* Known history of HIV infection or a known history of or is positive for Hepatitis B or Hepatitis C
* Presence of active infection requiring systemic therapy
* Corrected QT interval duration prolongation
* History of any one or more of the following cardiac conditions within the past 6 months: Cardiac angioplasty or stenting; Myocardial infarction; Unstable angina; History of Class III or IV congestive heart failure according to New York Heart Association classification
* History of cerebrovascular accident within the past 6 months
* Poorly controlled hypertension
* History of untreated deep venous thrombosis
* Presence of any non-healing wound, fracture, or ulcer, or presence of symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Recent hemoptysis
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Previous severe hypersensitivity reaction to another Monoclonal antibody. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the excipients in pazopanib tablets
* Has taken any prohibited medications that are listed in the protocol within 14 days of the first dose of study treatment. Subject has received or will receive a live vaccine within 30 days before the first administration of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-12-27 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs ) | From the start of study treatment (first dose) and, until the post-treatment follow-up visit (at least 30 days after the last dose of investigational product) for AEs, and until 90 days after last dose for SAEs
Part 1: To determine the dose limiting toxicity (DLT) and maximum tolerated regimen (MTR) | 8 weeks
  MTR is defined as the highest dose of pazopanib in combination with the highest dose of MK 3475 at which no more than 1 of 6 subjects experiences a DLT after a minimum of 8 weeks of treatment. DLT is defined as a drug-related AE starting in the first 8 weeks of treatment
Part 1: Number of subjects with permanent discontinuation of treatment, dose reductions, interruptions, or delays | 24 months
Part 1: Change from baseline in laboratory parameters | Average of 4 years
  Laboratory assessments include haematology, clinical chemistry, urine, coagulation and thyroid function test
Part 1: Change from baseline in vital signs | 30 days after the last dose of study treatment
  Vital sign measurements will include heart rate, temperature and blood pressure
Part 1: Change from baseline in cardiac parameters | 24 months
  Cardiac assessments will include Electrocardiogram (ECG) and Echocardiograms (ECHOs)
Part 1: Incidence and titer of anti MK 3475 antibodies | 24 months
  Subjects will be monitored for anti-MK 3475 antibodies throughout the study
Part 2: Progression-free survival (PFS) | Average of 4 years
  PFS is defined as the interval between the date of randomization and the earlier date of disease progression (using RECIST v1.1) or death due to any cause.

SECONDARY OUTCOMES:
Part 1: Dose escalation cohorts: pazopanib plasma concentrations and serum MK 3475 concentrations. | For Pazopanib: before and after the 1st and 2nd dose of MK-3475. For MK-3475: Until 6 months after the last dose of MK-3475
  For analysis of plasma pazopanib and serum MK 3475 concentrations, blood samples will be collected from all subjects
Part 1: Pharmacokinetic (PK) parameters in Expansion cohort | For Pazopanib: before and after the 1st and 2nd dose of MK-3475. For MK-3475: Until 6 months after the last dose of MK-3475
  Area under the plasma concentration-time curve from time 0 to 24 hrs (AUC[0-24], maximum observed concentration (Cmax), tmax, and concentration at 24 hours (C24) of pazopanib; Pre-dose (trough) concentration at the end of the dosing interval (Ctau), and apparent clearance following oral dosing CL/F of pazopanib will be determined if data permit.
Part 1 and Part 2: Overall response rate (ORR) | Average of 4 years
  Overall response rate is defined as the percentage of subjects, who achieved either a confirmed complete response (CR) or partial response (PR) by RECIST v1.1 and modified RECIST
Part 1 and Part 2: Clinical benefit rate | Average of 4 years
  Clinical benefit rate is defined as a confirmed response of CR or PR or at least 6-months stable disease by RECIST v1.1 and modified RECIST.
Part 1 and Part 2: Time to response | Average of 4 years
  Time to response is defined for all subjects with a confirmed CR or PR as per RECIST v1.1as the time from randomization until the first documented evidence of CR or PR (whichever status is recorded first)
Part 1 and Part 2: Duration of response | Average of 4 years
  Duration of response is defined for all subjects with confirmed CR or PR as the time from the first documented evidence of CR or PR until time of first documented disease progression or death due to any causes, whichever is first by RECIST v1.1 and modified RECIST
Part 2: PFS by modified RECIST | Average of 4 years
Part 1 and Part 2: Progression-free survival rate at 18 months (PFSR18) | 18 months
  PFSR18 will be calculated based on Kaplan-Meier estimates of Progression-free survival (PFS) at 18 months by RECIST v1.1 and modified RECIST
Part 2: Overall survival (OS) at 18 months | 18 months
  Overall survival at 18 months will be summarized based on the Kaplan-Meier method.
Part 2: Overall survival (OS) | Average of 4 years
  Overall survival will be summarized using Kaplan-Meier survival curves
Part 2: Incidence and severity of AEs and SAEs | From the start of study treatment (first dose) and, until the post-treatment follow-up visit (at least 30 days after the last dose of investigational product) for AEs, and until 90 days after last dose for SAEs
Part 2: Number of subjects with permanent discontinuation of treatment, dose reductions, interruptions, or delays | Average of 4 years
Part 2: Change from baseline in laboratory parameters | Average of 4 years
  Laboratory assessments include haematology, clinical chemistry, urine, coagulation and thyroid function test
Part 2: Change from baseline in vital signs | Average of 4 years
  Vital sign measurements will include heart rate, temperature and blood pressure
Part 2: Change from baseline in cardiac parameters | Average of 4 years
  Cardiac assessments will include ECG and ECHOs
Part 2: Incidence and titer of anti MK 3475 antibodies in patients treated with pazopanib + MK 3475 and single-agent MK 3475 | Until 6 months after the last dose of MK-3475
  Subjects will be monitored for anti-MK 3475 antibodies throughout the study
Part 2: PK parameters in randomized phase | For Pazopanib: Until Dose 49 of MK-3475.
  For analysis of plasma pazopanib and serum MK 3475 concentrations, blood samples will be collected from all subjects. AUC[0-24], Cmax, tmax, and C24 of pazopanib alone and in combination with MK 3475; Cmax, Ctau, and apparent clearance following oral dosing CL/F of pazopanib will be determined if data permit.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (3):
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Nashville, Tennessee
- United Kingdom (2):
  - Novartis Investigative Site, Manchester, Lancashire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com